CLINICAL TRIAL: NCT07311512
Title: The Effect of Professional Mechanical Plaque Removal (PMPR) and Chlorhexidine Mouthwash on Salivary and Acquired Enamel Pellicle (AEP) Proteins and Vascular Function and Inflammation in People With Periodontal Disease
Brief Title: PMPR and Chlorhexidine on Periodontal Disease and Vascular Function
Acronym: CHX-PMPR-PERIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahdi Mutahar (Other)
Collaborators: Loughborough University (Other); Temple University (Other); Imperial College London (Other)
Responsible Party: Sponsor-Investigator, Mahdi Mutahar, Dr. Mahdi Mutahar, University of Portsmouth
Organization: University of Portsmouth (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS Project ID: 351521; REC reference: 25/WA/0160 (Other: National Health Service, Wales Research Ethics Committee 6)
Record Dates: First submitted 2025-11-14; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Disease (PD); Cardio Vascular Disease; Oral-Systemic Link; Vascular Dysfunction; Endothelial Function and Arterial Stiffness
Keywords: Chlorhexidine Mouthwash; Periodontal Disease; Professional Mechanical Plaque Removal (PMPR); Salivary Proteins; Acquired Enamel Pellicle (AEP); Proteomics; Vascular Function; Endothelial Function; Flow-Mediated Dilation (FMD); Pulse Wave Analysis (PWA); Pulse Wave Velocity (PWV); Blood Pressure; Nitric Oxide; Nitrate reducing bacteria (NRB); Inflammation biomarkers; Oral-Systemic Link; Saliva Collection; Blood Sample Collection; Cardiac Output
MeSH Terms: conditions — Periodontal Diseases | interventions — Chlorhexidine; Mouthwashes

STUDY DESIGN:
Intervention Model Description: * Participants will be identified by School of Dental Health and Care Professions (SDHCP) dental clinicians and research team.Participants will be provided study information ≥24h before appointments. After consent, periodontal screening per BSP 2017 guidelines will be conducted by the calibrated dental clinicians.
  * Eligible participants will complete medical/dental history, saliva and AEP sampling at SDHCP. Vascular assessments will be performed at the School of Psychology, Sport and Health Sciences (SPSHS) using iontophoresis, flow-mediated dilation, pulse wave velocity, cardiac output , blood pressure, and blood sample collection.
  * PMPR will be done once at baseline (Visit 1) as standard care by the dental clinicians at SDHCP with research procedures performed before and after the PMPR procedure.
  * At Visit 2, participants will be randomised to receive either 0.2% chlorhexidine or placebo mouthwash (10 ml, 1 min, twice daily, 14 days), with follow-up at Day 1, Day 14, and Day 90.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMPR + Placebo (Placebo Comparator): Arm 2 - Participants in this arm will receive PMPR using ultrasonic scalers at baseline (Visit 1) as part of routine care. At Visit 2 (Day 1), participants will be randomised to receive a placebo mouthwash, identical in taste, color, appearance to the chlorhexidine mouthwash.
  - This placebo comparator will allow assessment of the effect of chlorhexidine versus no active antibacterial treatment, while keeping participants and researchers blinded. Participants follow the same regimen (10 ml rinse, 1 min, twice daily for 14 days), with saliva, AEP, blood, and vascular function measurements collected at baseline, Day 1, Day 14, and Day 90.
  Interventions: Other: Placebo mouthwash
- PMPR + CHX (Active Comparator): * Arm 1
  * Participants in this arm will receive PMPR using ultrasonic scalers at baseline (Visit 1), as part of their standard care. At Visit 2 (Day 1), they will be randomised to receive 0.2% chlorhexidine mouthwash (10 ml, 1 min, twice daily for 14 days), with saliva, Acquired Enamel Pellicle (AEP), blood sample collection, and vascular function measurements done at baseline(Day 0), Day 1, Day 14, and Day 90.
  Interventions: Other: Chlorhexidine (0.2%) mouthwash

INTERVENTIONS:
Other: Chlorhexidine (0.2%) mouthwash — PMPR is a routine standard dental treatment for gingivitis and PD, and will not form part of the research intervention. The research intervention consists of using 0.2% chlorhexidine mouthwash (10 ml, rinsed for 1 minute, twice daily for 14 days).
  Other Names: Chlorhexidine Mouthwash
  Arms: PMPR + CHX
Other: Placebo mouthwash — PMPR is a routine standard dental treatment for gingivitis and PD, and will not form part of the research intervention. The research intervention consists of a placebo mouthwash (10 ml, 1 min, twice daily for 14 days). The placebo mouthwash (control) is designed to resemble commercially available products but without the active ingredient. Use of this has been ethically approved (IRAS Project ID: 333173), validated and tested in the investigator's previous studies (Data to be published).
  Arms: PMPR + Placebo

SUMMARY:
* Gum inflammation is called gingivitis. Gum disease, known as periodontal disease, is a long-term inflammation of the gums and bone around teeth, leading to tooth loss. Both gingivitis and periodontal disease are also linked to other health problems, including heart disease. Additionally, salivary proteins play a role in maintaining oral health. For example, a protective layer called the salivary pellicle (SP) forms on teeth after tooth brushing and helps defend against harmful bacteria.
* Nitrate-reducing bacteria (NRB) are also present in saliva and play a role in oral and cardiovascular health by converting nitrate to nitric oxide (NO). This compound supports blood vessel health and overall cardiovascular function. Therefore, NRB's abundance is linked to lower blood pressure and improved cardiovascular health.
* Standard treatments for gum disease include deep cleaning (also called professional mechanical plaque removal, or PMPR), and sometimes chlorhexidine (CHX) mouthwash is used with PMPR to help reduce mouth bacteria. However, while CHX is effective against plaque (a sticky film of bacteria on the tooth surface), it may reduce the activity of "nitrate-reducing" bacteria (NRB), which are important for producing nitric oxide (NO).
* This study investigates the impact of deep cleaning (PMPR) with and without Chlorhexidine mouthwash on salivary and SP proteins, as well as blood vessel function, in people who have gum disease. By examining these links, the investigators aim to gain a deeper understanding of how oral care practices may impact overall health, particularly heart health.

DETAILED DESCRIPTION:
* **Introduction**

  * Periodontal disease (PD) is a chronic inflammatory condition affecting the tissues supporting teeth, including gums, bone, and ligaments, and is associated with a 19% increased risk of cardiovascular disease. It starts with gum inflammation, known as gingivitis. Both chronic gingivitis and PD have multiple causes including poor oral hygiene, smoking, diabetes, genetics, stress, age, and certain medications, and PD contributes significantly to healthcare costs ($54 billion direct, $25 billion indirect annually).
  * The key approach for managing PD is non-surgical, typically involving Professional Mechanical Plaque Removal (PMPR), with or without adjunct antiseptic mouthwashes such as 0.2% chlorhexidine (CHX). While CHX is effective in reducing dental plaque, concerns exist regarding its impact on beneficial oral nitrate-reducing bacteria (NRB), which play a critical role in systemic nitric oxide (NO) pathways and cardiovascular homeostasis. Altering the oral microbiome may influence vascular function, including blood pressure and endothelial health.
  * This study investigates the effects of PMPR, performed as standard periodontal therapy, and adjunctive CHX mouthwash on salivary and acquired enamel pellicle (AEP) proteins, oral microbiome, NRB activity, and vascular function in individuals with PD.
* **Study Design Overview**
* A total of 30 adult participants with clinically confirmed gingivitis and/or periodontal disease will be enrolled and followed at four assessment points over a three-month period.
* Recruitment Process and Practicalities

Under the supervision of the academic supervisor, potential research participants will be recruited via the following steps:

* Research participants recruited from SDHCP dental clinics:

  * Step 1: Providing Study Information to Potential Participants Clinicians at the University of Portsmouth (SDHCP), Dr. Anish Patel, Prof. Chris Louca, and Dr. Bhavin Dedhia, will inform patients about the study during their routine clinical appointments. Study materials, including the Participant Information Sheet and Invitation Letter, will be provided at least 24 hours before the first appointment, allowing individuals time to consider participation.
  * Step 2: Participant Follow-Up Participants who wish to volunteer for the study will then be contacted by the research team. The PhD researcher will explain the study in more detail, answer any questions, and confirm their willingness to participate. This process ensures that participants have at least 24 hours to consider their involvement before their appointment. The consent form will be signed by the individuals in person, before their oral screening, on their first visit.
  * Eligibility Screening: Consented participants will undergo a routine clinical examination by the clinicians using the standard British Society of Periodontology (BSP) 2017 classification, focusing on individuals with BPE codes 1 to 4 for gingivitis and subsequent diagnosis of periodontitis (stages 1 and 2).
* Research participants recruited from community centres:

  -- Step 1: Providing Study Information to Potential Participants: The PhD researcher will engage with the public by visiting community centres in Portsmouth and delivering informational talks about the study. Study materials, including the Participant Information Sheet and Invitation Letter, will be provided to allow potential participants at least 24 hours before their first appointment.
  * Step 2: Participant Follow-Up Interested individuals will be contacted by the research team to review the study participant information sheet (PIS), address any questions, and confirm their willingness to participate. Eligible participants will then be invited to the University of Portsmouth SDHCP dental clinics to receive routine dental treatment, which will include participation in the research study.
  * After screening and completion of questionnaires and forms, participants will be matched based on factors that may affect salivary proteins at baseline, including age (30-75 years), smoking status, BPE gingival score, periodontal disease classification, clinical severity of caries, dental erosion, and presence of diabetes.
  * The study will be composed of two sequential phases:
  * (i) Observational phase: Measure changes in salivary and Acquired Enamel Pellicle (AEP) or salivary pellicle (SP) protein composition and vascular function before and after routine PMPR.
  * (ii) Randomised, double-blind, placebo-controlled interventional phase: Participants will receive either CHX mouthwash or placebo mouthwash for two weeks following PMPR to evaluate combined or isolated effects on oral and vascular parameters.
  * Unstimulated whole mouth saliva (WMS) and AEP samples will be collected at baseline (Day 0), Day 1, Day 14, and Day 90. Proteomic and protein quantification techniques will map changes in both host and bacterial proteins. DNA-based microbiome analysis (16S rRNA sequencing) will examine shifts in bacterial composition, with particular attention to NRB and periodontal pathogens.
  * Vascular Function Assessments will include:
  * (i) Flow-Mediated Dilation (FMD): Large blood vessel endothelial function (ultrasound)
  * (ii) Pulse Wave Analysis (PWA) and Pulse Wave Velocity (PWV): Arterial stiffness
  * (iii) Iontophoresis: Small blood vessel endothelial function
  * (iv) Cardiac Output: The volume of blood pumped by the heart into the systemic circulation per minute, will be measured using PhysioFlow
  * (v) Blood Pressure: Including Mean Arterial Pressure (MAP)
  * (vi) Blood samples: Inflammatory plasma biomarkers (IL-6, IL-10, TNF-alpha)
* **Power and Sample Size Calculations**

  * (i) Observational phase: N = 6, paired t-test, effect size 0.87, 80% power, α < 0.05
  * (ii) Interventional phase: Based on salivary biomarker MMP-8. ANOVA repeated measures with 90% power, α < 0.05, effect size f = 0.87, requiring 12 participants per group. Accounting for 14% dropout, n = 15 per group, total N = 30.
  * Standardised procedures, examiner calibration, identical toothpaste and mouthwash containers, and allocation concealment will minimise bias and variability.
  * Participant Materials Key study documents, such as the participant information sheet and consent form, were shared with the PPI group for review. They provided explicit feedback on the clarity and accessibility of these materials, resulting in revisions to ensure the language is easy to understand and free of jargon. This has made the study more approachable for potential participants.
* **Storage of Data**

  -- No identifiable personal data will be published. All data will be linked-anonymised. Results published in journals or data repositories will contain only anonymised data.
* **Analysis of Data**

  * i) Saliva Proteomics Analysis - Samples generated at School of Dental, Health and Care Professions (SDHCP), University of Portsmouth; proteomics analysis at Imperial College London. Saliva samples will be analysed for changes in salivary proteins, using Perseus software (Perseus_v2.1.3.0.zip), run on .NET Desktop Runtime.
  * ii) Saliva Oral Microbiome Analysis - Samples generated at SDHCP, analysed at Temple University, USA, using Next-generation sequencing methods.
  * iii) Acquired Enamel Pellicle Proteins - Analysed using SDS-PAGE and Western blotting.
  * iv) Nitrate-Reducing Bacteria Activity - Generated at SDHCP, analysed at Loughborough University.
  * v) Vascular Function Data - Generated and analysed at School of Psychology, Sport and Health Sciences (SPSHS), University of Portsmouth.
* **Clinical Significance**

  --This study will reveal how PMPR and adjunctive CHX mouthwash modulate the oral proteome and microbiome, and how these changes relate to vascular function. Findings will clarify the systemic effects of commonly used oral antiseptics, particularly on NRB and vascular function. Results will inform best practices for periodontal therapy, shaping future oral and systemic health guidelines.
* **Dissemination**

The findings from this study will be disseminated through multiple channels:

* (i) Peer-reviewed journals: Results will be submitted to high-impact dental, oral health, and cardiovascular journals.
* (ii) Scientific conferences: Findings will be presented at national and international conferences in periodontology, dentistry, and vascular research.
* (iii) Public engagement: Lay summaries will be made available to participants and the public via the University of Portsmouth website and social media platforms.
* (iv) Data sharing: De-identified datasets and analytical methods may be shared with other researchers upon reasonable request, following ethical approval and data protection guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a minimum of 2 natural teeth in each sextant (at least 12 teeth overall).
* Individuals with clinically diagnosed gingivitis and/or early periodontitis (stage 1 and 2)
* Must not have undergone periodontal maintenance therapy (PMPR) within the last 6 months.
* Must not currently be wearing orthodontic appliances, due to their effect on oral microbiota and plaque composition.
* Must not be using removable orthodontic appliances, as they increase plaque accumulation.
* Must not have taken any antibiotic treatments within the last 3 months.
* Must be able to provide written informed consent.
* Individuals with dental erosion or caries will still be included but matched during the baseline visit.

Exclusion Criteria:

* Individuals under regular medication within one month of the study start date for any medical condition (such as hypertension and/or diabetes)
* Pregnant or breastfeeding individuals.
* Individuals requiring an interpreter or who are non-English speakers.
* Individuals unable to provide written informed consent.
* Individuals participating in another ongoing clinical study (other than observational studies) within 3 months prior to or during this study.
* Individuals who have used mouthwash or tongue scrapers in the last 6 weeks.
* Individuals who consume 20 or more cigarettes per day.
* Individuals who consume more than 5 alcoholic drinks per day.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Proteomics - Salivary Protein Analysis | Analysed for WMS samples collected on Day 0, Day 1, Day 14, and Day 90.
  Purpose: To identify inflammatory and protective proteins, monitor changes post-PMPR in saliva.
  * Method ( Protocol from Imperial College, London):
  * Reduction & Alkylation: A 10 μL aliquot of saliva will be thawed and mixed with 7 μL of ammonium bicarbonate buffer on ice. For reduction and alkylation, 5 μL each of TCEP and CAA will be added, maintaining a pH of 7-8 to ensure proper modification of disulfide bonds and cysteine residues.
  * SP4 Protocol: Following reduction and alkylation, the SP4 protocol will be implemented by adding 80 μL of LC/MS-grade acetonitrile to precipitate proteins; the mixture will be centrifuged to separate the supernatant, and the pellet will be washed three times with ethanol for thorough purification.
  * Digestion: The purified pellet will then be resuspended in stock trypsin by adding 20 μL 25 mM ammonium bicarbonate to lyophilised powdered trypsin (powdered sequencing grade modified trypsin) and incubate overnight at 37°C, and incubated overnight.

SECONDARY OUTCOMES:
Salivary Flow-Rate | Day 0, Day 1, Day 14, and Day 90
  - Unstimulated whole mouth saliva (uWMS) sample will be used to measure salivary flow rate. Salivary flow rate (mL/min) is calculated as:
  Salivary flow rate (mL/min) = (Weight of tube with saliva - Weight of empty tube) ÷ Collection time (min).
Salivary pH | Day 0, Day 1, Day 14, and Day 90
  * An unstimulated whole mouth saliva (uWMS) sample will be used to measure salivary pH.
  * Following saliva collection, salivary pH will be measured using a single-electrode digital pH meter (Lutron Electronic Enterprise Co., Ltd., Model PH-208, Taiwan).
Oral Microbial Composition | Day 0, Day 1, Day 14, and Day 90
  * Microbial composition of the saliva will be characterised by DNA extraction and 16S rRNA sequencing to observe oral microbiome shifts following PMPR.-
  * Purpose: To characterise oral microbiome shifts after PMPR.
  * Method/techniques: DNA extraction; 16S rRNA sequencing.
  * Bacterial genomic DNA will be extracted from WMS and AEP samples using standard methods or commercial kits. The extracted DNA will serve as the template for PCR amplification of 16S rRNA gene fragments (500-1,500 bp). - Prepared saliva and pellicle samples will be sent to the Oral Microbiome Research Laboratory at Temple University (USA) for DNA extraction and 16S rRNA sequencing, with a Material Transfer Agreement (MTA) in place. - Microbial DNA will be extracted from 1-3 mL of samples using Qiagen QIAamp or Vazyme VAMNE kits. DNA quantification will be performed using fluorometric methods (Qubit), and purity will be assessed by absorbance. Three sterile water blanks will be included as controls.
Acquired Enamel Pellicle (AEP) Protein Composition | Day 0, Day 1, Day 14, Day 90
  - Protein profile will be assessed in AEP. The purpose is to understand tooth-surface protective vs. pathogenic protein changes. Pellicle will be collected using filter strips; protein elution and analysis.
  Parameters Assessed: Structural and functional protein variations (such as- albumin, cystatins, mucins, PRPs). - Purpose: To detect and compare key structural protein changes across study time points. - Methods/techniques: SDS-PAGE and Western blot. Sodium dodecyl sulfate-polyacrylamide gel electrophoresis (SDS-PAGE) is a discontinuous electrophoresis method commonly used to separate proteins with molecular weights between 5 and 250 kDa. SDS acts as a surfactant, masking the proteins' natural charges and giving them nearly identical charge-to-mass ratios. Under a constant electric field, proteins migrate toward the anode at speeds determined by their mass, allowing accurate size-based separation.Western blot is a molecular technique used to detect and quantify specific proteins
Nitrate Reducing Activity of the Oral Bacteria | Analysed for the nitrate rinse samples collected on Day 0, Day 1, Day 14, and Day 90.
  * Purpose: To evaluate the oral microbiota's nitrate-reducing capacity.
  * To evaluate bacterial role in nitric oxide pathways.
  * Method: Nitrate rinse; incubation; centrifugation; nitrite quantification.
  To assess nitrate-reducing activity in WMS samples, a stock solution will be prepared by dissolving 1011 mg potassium nitrate in 1 L of ultrapure water. Aliquots of 10 mL will be stored in 15 mL Falcon tubes at -20°C until use.
  * For the procedure, one aliquot will be thawed and used as a rinse solution. Participants will rinse their mouths with 10 mL of the solution for 5 minutes under timed supervision. The expectorated rinse will be collected in a 50 mL Falcon tube and transferred into microcentrifuge tubes.
  * Samples will be centrifuged at 10,000 rpm for 10 minutes. The supernatant will be collected, transferred into a new tube, and stored at -20°C for later analysis of nitrite concentration.
Flow-Mediated Dilation (FMD)- Large Blood Vessel Endothelial Function Test (Ultrasound) | On Day 0, upon participant arrival at the first visit, prior to PMPR treatment. On Day 1, i.e. 24 hours after PMPR treatment. On Day 14, two weeks following chlorhexidine/placebo mouthwash use, and then on Day 90, three months post-PMPR treatment.
  * Brachial artery FMD will be used to assess endothelial function following a 5-minute ischemic stimulus induced by forearm cuff inflation. Measurements will be performed in the supine position on the right arm, with the cuff placed distal to the olecranon process.
  * A 12-MHz linear array ultrasound probe will be used to image the brachial artery while simultaneously recording B-mode images and Doppler blood velocity traces. Depth, focus, and gain settings will remain consistent, and the transducer location will be documented for reproducibility.
  * After a 60-second baseline, the cuff will be inflated to 220 mmHg for 5 minutes. Ultrasound recordings will continue during inflation and for 3 minutes post-deflation. All scans will be performed by the same researcher for each participant.
  * Brachial artery diameter, blood flow, and shear rate will be analysed using automated edge-detection and wall-tracking software to minimise investigator bias.
Iontophoresis- Small Blood Vessel Endothelial Function Test | On Day 0, upon participant arrival at the first visit, prior to PMPR treatment. On Day 1, i.e. 24 hours after PMPR treatment. On Day 14, two weeks following chlorhexidine/placebo mouthwash use, and then on Day 90, three months post-PMPR treatment.
  * Iontophoresis will be used to assess microvascular endothelial function through transdermal drug delivery with a low-intensity electric current. Participants will acclimatize for 30 minutes in a room maintained at 23°C before receiving acetylcholine (ACh, 1%) and sodium nitroprusside (SNP, 0.01%) on the volar forearm.
  * The skin will be cleaned with water for injection, and two perspex rings will be placed as anode and cathode, connected to the iontophoresis controller. Each chamber will contain 0.5 mL of drug solution. The stimulation protocol will include four pulses at 25 μA, followed by single pulses at 50, 100, 150, and 200 μA, each lasting 20 seconds with 120-second intervals.
  * Skin blood flow will be measured using Laser Doppler probes connected to a perfusion monitor, with data recorded via PowerLab and LabChart software. Cutaneous vascular conductance (CVC) will be calculated as skin flux/MAP.
Cardiac Output (CO) | On Day 0, upon participant arrival at the first visit, prior to PMPR treatment. On Day 1, i.e. 24 hours after PMPR treatment. On Day 14, two weeks following chlorhexidine/placebo mouthwash use, and then on Day 90, three months post-PMPR treatment.
  * Cardiac output (CO) will be measured noninvasively using the Physio Flow PF-05 Lab1 device with thoracic electrode placement. Two electrodes placed at the sternal manubrium and lower thorax will monitor EKG for heart rate, while four electrodes at the neck base and xiphoid process will measure impedance signals.
  * Skin will be prepared by shaving and cleaning to optimise signal quality. For participants with pacemakers, neck electrodes will be positioned opposite the device. Calibration will be performed by acquiring stable signals over 30 heartbeats with simultaneous blood pressure measurement.
  * The system will provide heart rate, stroke volume, CO, and other hemodynamic parameters, with data reviewed and stored for analysis.
Pulse Wave Analysis (PWA) | On Day 0, upon participant arrival at the first visit, prior to PMPR treatment. On Day 1, i.e. 24 hours after PMPR treatment. On Day 14, two weeks following chlorhexidine/placebo mouthwash use, and then on Day 90, three months post-PMPR treatment.
  - Pulse Wave Analysis (PWA) will be performed to assess central aortic hemodynamic parameters. After a 5-minute rest, brachial pressure waveforms will be recorded and used to derive aortic waveforms via a transfer function. Output will include pulse pressure (PP), augmentation pressure (AP), and augmentation index (AI75). Results will be displayed graphically and compared with population norms using the SphygmoCor XCEL system.
Pulse Wave Velocity (PWV) | On Day 0, upon participant arrival at the first visit, prior to PMPR treatment. On Day 1, i.e. 24 hours after PMPR treatment. On Day 14, two weeks following chlorhexidine/placebo mouthwash use, and then on Day 90, three months post-PMPR treatment.
  - Pulse Wave Velocity (PWV) will be measured as an index of arterial stiffness. Participants will rest in the supine position for 5 minutes before measurement. A femoral cuff will be placed on the thigh, and carotid pressure will be recorded with a tonometer to calculate transit time and derive PWV in m/s. Results will be compared with population data.
Salivary Nitrite Concentration | Day 0, Day 1, Day 14, and Day 90.
  * Ozone-based chemiluminescence, a biochemical test, will be used to measure nitric oxide (NO) metabolites, primarily nitrite (NO₂-), in saliva samples. In this method, NO reacts with ozone to produce an excited form of nitrogen dioxide, which is detected as a chemiluminescent signal.
  * Saliva samples will be analysed for nitrite concentrations using a Sievers nitric oxide analyser (Sievers NOA 280i).
Salivary Nitrate Concentration | Day 0, Day 1, Day 14, and Day 90.
  * Ozone-based chemiluminescence, a biochemical test, will be used to measure nitric oxide (NO) metabolites, such as nitrate (NO₃-), in saliva samples. In this method, NO reacts with ozone to produce an excited form of nitrogen dioxide, which is detected as a chemiluminescent signal.
  * Saliva samples will be analysed for nitrate concentrations using a Sievers nitric oxide analyser (Sievers NOA 280i).
Plasma Nitrite Concentration | Day 0, Day 1, Day 14, and Day 90
  - Plasma nitrite (NO₂-) levels will be quantified using ozone-based chemiluminescence. In this method, nitric oxide reacts with ozone to generate excited nitrogen dioxide, producing a measurable chemiluminescent signal. Plasma samples will be centrifuged and stored at -80 °C until analysis with a Sievers Nitric Oxide Analyser (NOA 280i)
Plasma Nitrate Concentration | Day 0, Day 1, Day 14, and Day 90
  - Plasma nitrate (NO₃-) levels will be quantified using ozone-based chemiluminescence. In this method, nitric oxide reacts with ozone to generate excited nitrogen dioxide, producing a measurable chemiluminescent signal. Plasma samples will be centrifuged and stored at -80 °C until analysis with a Sievers Nitric Oxide Analyser (NOA 280i)
Blood Pressure (BP) | On Day 0, upon participant arrival at the first visit, prior to PMPR treatment. On Day 1, i.e. 24 hours after PMPR treatment. On Day 14, two weeks following chlorhexidine/placebo mouthwash use, and then on Day 90, three months post-PMPR treatment.
  * Blood pressure in the brachial artery will be measured after 30 minutes of seated rest in a quiet room, using an automated sphygmomanometer. Five consecutive readings will be taken, with a 1-minute rest between each measurement.
  * The average of three readings will be recorded, including the mean values for SBP, DBP, and MAP.
Inflammatory Biomarkers in Blood | Analysed for the venous blood samples collected on Day 0, Day 1, Day 14, and Day 90.
  * Enzyme-Linked Immunosorbent Assay (ELISA) Duoset kits will be used to quantify blood biomarkers, including IL-6, IL-10, and TNFα, and to assess systemic inflammation and its association with periodontal disease and vascular function. The kits use a sandwich ELISA approach, with a capture antibody pre-coated onto a microplate, followed by sample application.
  * This method allows precise measurement of cytokines and acute-phase proteins from participants' blood samples. High specificity and sensitivity enable detection of both pro-inflammatory (IL-6, TNFα) and anti-inflammatory (IL-10) markers. Results will provide insights into the inflammatory response and its modulation before and after PMPR treatment.
Efficacy of PMPR ± CHX Mouthwash on Bleeding on Probing (Periodontal Clinical Index) | Day 0, Day 1, Day 14, Day 90
  To evaluate and assess the efficacy of Periodontal Mechanical Plaque Removal (PMPR) combined with 0.2% CHX mouthwash on Bleeding on Probing (BoP)
  * BOP will be recorded at six sites per tooth as: 0 (minimum) = no bleeding, 1 (maximum) = bleeding on probing.
  * Scores will be expressed as the percentage of bleeding sites per participant, with a minimum to maximum range (0-100%).
  * Lower scores indicate a better periodontal outcome; a reduction reflects improvement following PMPR ± CHX mouthwash.
  * This outcome will assess the short-term clinical efficacy of CHX mouthwash adjunctive to PMPR in individuals with periodontal disease.
Efficacy of PMPR ± CHX Mouthwash on Probing Pocket Depth (Periodontal Clinical Index) | Day 0, Day 1, Day 14, Day 90
  To evaluate and assess the efficacy of Periodontal Mechanical Plaque Removal (PMPR) combined with 0.2% CHX mouthwash on Probing Pocket Depth (PPD)
  * PPD will be measured in millimetres at six sites per tooth and categorised as: 0 (minimum) = ≤3 mm, 1 = 4-5 mm, 2 (maximum)= ≥6 mm. Lower scores indicate a better periodontal outcome. - Efficacy will be assessed as mean change in PPD (mm) and as percentage of pocket closure, defined as sites with baseline PPD ≥4 mm reducing to ≤3 mm at follow-up.
  * This outcome will assess the short-term clinical efficacy of CHX mouthwash adjunctive to PMPR in individuals with periodontal disease.
Efficacy of PMPR ± CHX Mouthwash on Clinical Attachment Level (Periodontal Clinical Index) | Day 0, Day 1, Day 14, Day 90
  To evaluate and assess the efficacy of Periodontal Mechanical Plaque Removal (PMPR) combined with 0.2% CHX mouthwash on the Clinical Attachment Level (CAL)
  * Clinical Attachment Level (CAL) will be calculated by combining probing pocket depth and gingival recession measurements.
  * CAL will be measured in millimetres at six sites per tooth and categorised as: 0 (minimum) = 0-2 mm, 1 = 3-4 mm, 2 (maximum) = ≥5 mm.
  * The mean change in CAL (mm) will then be compared between the two groups (PMPR + CHX vs. PMPR + placebo).
  * Lower scores indicate a better periodontal outcome; a reduction reflects attachment gain following use of PMPR ± CHX mouthwash.
  * This index will be used to assess the short-term clinical efficacy of CHX mouthwash, adjunctive to PMPR, in individuals with periodontal disease.
Efficacy of PMPR ± CHX Mouthwash on Plaque Index | Day 0, Day 1, Day 14, Day 90
  To evaluate and assess the efficacy of Periodontal Mechanical Plaque Removal (PMPR) combined with 0.2% CHX mouthwash on Plaque index (PI).
  * A score of 0,1,2,3,4,5 will be used to record the PI on the buccal and lingual surfaces of the teeth (except third molars) using the Turesky-modified scoring criteria.
  * Scoring system:
  * 0 (minimum)= No plaque; 1 = flecks at cervical margin; 2 = thin band ≤1 mm; 3 = band >1 mm covering <⅓ surface; 4 = plaque covering ≥⅓-<⅔; 5 (maximum)= plaque covering ≥⅔ of the surface.
  * Scores will be averaged across all surfaces to obtain a mean PI score from minimum to maximum, with a range of 0-5.
  * Lower scores indicate better oral hygiene; a reduction reflects improvement following PMPR ± CHX mouthwash.
  * This index will be used to assess the short-term clinical efficacy of CHX mouthwash, adjunctive to PMPR, in individuals with periodontal disease.
Efficacy of PMPR ± CHX Mouthwash on Gingival Index | Day 0, Day 1, Day 14, Day 90
  To evaluate and assess the efficacy of Periodontal Mechanical Plaque Removal (PMPR) combined with 0.2% CHX mouthwash on Löe & Silness Gingival Index (GI).
  * GI will be assessed at four sites per tooth (mesial, distal, buccal, lingual) and scored (on a minimum 0 to a maximum 3) with: 0 = normal, 1 = mild inflammation, 2 = moderate inflammation, 3 = severe inflammation. Scores will be averaged across all sites to give a mean GI score (range 0-3). Lower scores indicate better gingival health; a reduction reflects improvement following PMPR ± 0.2% CHX mouthwash.
  * Gingivitis severity classification:
  * Mild gingivitis: 0.1-1.0; Moderate gingivitis: 1.1-2.0; Severe: 2.1-3.0
  * This index will be used to assess the short-term clinical efficacy of CHX mouthwash on GI, adjunctive to PMPR, in individuals with periodontal disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD, but summary-level results will be disseminated through peer-reviewed publications and conference presentations.

REFERENCES:
- See also: Dr. Mahdi Mutahar, Senior Lecturer at the University of Portsmouth Dental Academy, supervises Saagarika Sharma's PhD project on the effect of PMPR and chlorhexidine mouthwash on salivary, pellicle proteins and vascular function. — https://www.port.ac.uk/about-us/structure-and-governance/our-people/our-staff/mahdi-mutahar
- See also: This University of Portsmouth project investigates how professional mechanical plaque removal and chlorhexidine mouthwash affect salivary proteins, acquired enamel pellicle and vascular function in individuals with periodontal disease. — https://researchportal.port.ac.uk/en/projects/the-effect-of-pmpr-and-chlorhexidine-mouthwash-on-salivary-and-ac

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Procedure and Statistical Test Analysis (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT07311512/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Power Calculation (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT07311512/Prot_SAP_001.pdf
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT07311512/ICF_002.pdf